CLINICAL TRIAL: NCT04977076
Title: Comparison Between Direct Oral Anticoagulation (DOAC) Interruption and DOAC Continuation in Patients Undergoing Elective Invasive Coronary Angiography or Percutaneous Coronary Intervention
Acronym: SLIM-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: METCZ20210099
Record Dates: First submitted 2021-07-20; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, 1:1 randomized, investigator initiated study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupted NOAC use (group 1) (Active Comparator): Patients in group 1 will receive standard care. Therefore, DOAC use will be interrupted at least 24 hours in advance of ICA or PCI. Based on the renal clearance, last DOAC intake may be extended to 48 hours prior to the procedure [Table 2]. After the procedure, patients will continue using their DOAC as usual.
  Interventions: Other: Interrupted NOAC use
- Uninterrupted NOAC use (group 2) (Experimental): In group 2, all patients will continue to use their specific DOAC as usual. This means that no adjustments of DOAC use will be made before and after ICA or PCI. After the procedure patients will continue to use DOAC from the next planned dose.
  Interventions: Other: Uninterrupted NOAC use

INTERVENTIONS:
Other: Uninterrupted NOAC use — Continuing NOAC use in advance of elective CAG or PCI.
  Arms: Uninterrupted NOAC use (group 2)
Other: Interrupted NOAC use — Usual care, interruption of NOAC prior to procedure.
  Arms: Interrupted NOAC use (group 1)

SUMMARY:
A prospective, multicenter, 1:1 randomized, investigator initiated study. Goal of this study is to examine the safety of uninterrupted periprocedural NOAC use.

DETAILED DESCRIPTION:
Rationale: Patients with atrial fibrillation (AF) often have coexisting coronary artery disease (CAD). An estimated 5 to 15% of all AF patients will require coronary stenting. Direct Oral Anticoagulants (DOAC) are more commonly used in preventing thromboembolic complications in patients with AF, thereby substituting the use of Vitamin-K Antagonists (VKA). Therefore, many patients undergoing invasive coronary angiography (ICA) and percutaneous coronary intervention (PCI) are taking direct oral anticoagulants (DOAC). In patients using VKA it is recommended to defer elective coronary angiography until INR is <2.2 when radial artery access is used. However, no large clinical trials have proven the safety of continuing DOAC use when undergoing ICA or PCI. The current guidelines recommend interrupting DOAC treatment at least 24 before ICA or PCI; however, this recommendation is only based on limited data. Clinical decisions on DOAC use must therefore be based on clinical trials in which substantial numbers of patients with Acute Coronary Syndrome (ACS) were included.

Objective: To study the safety of DOAC continuation in patients undergoing ICA or PCI.

Study design: A prospective, multicenter, 1:1 randomized, investigator initiated study.

Study population: Patients aged >18 years using DOAC and undergoing elective ICA or PCI.

Intervention: The intervention group will continue using DOAC as usual. No adjustments of DOAC use will be made before and after ICA or PCI. The control group will receive standard care. DOAC use will be interrupted at least 24-48 hours in advance of ICA or PCI, based on renal clearance and DOAC specimen.

Main study parameters/endpoints: : Non-CABG related in-hospital major bleeding (BARC 3 or 5).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Only a small burden is associated with participation. Patients are asked to fill out a questionnaire after 30 days. Patients in the control group may have a mildly higher risk of thromboembolic complications and patients in the intervention group may have a mildly higher risk of bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years using DOAC and undergoing elective ICA or PCI.
* Provided signed informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

Any of the following:

* Patients initially presenting with Acute Coronary Syndrome (STEMI, NSTEMI, UA)
* Patients <18 years old
* Calculated CLCR <30 mL/min
* Patients simultaneously participating in another clinical trial
* History or condition associated with increased bleeding risk, as listed below:

  * Major surgical procedure within 30 days before the procedure
  * Known inaccessible radial artery during previous procedure
  * History of GI bleeding in the previous 6 months
  * History of intracranial, intraocular, spinal, or atraumatic intra-articular bleeding
  * Chronic bleeding disorder
  * Known intracranial neoplasm, arteriovenous malformation, or aneurysm
  * Known anemia with last measured haemoglobin value <6 mmol/L [9.67 g/dL]
  * Current pregnancy or breast-feeding
  * Known significant liver disease (e.g., acute clinical hepatitis, chronic active hepatitis, cirrhosis), or ALT >3 x the ULN
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1214 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Bleeding | 30 days
  Non-CABG related in-hospital major bleeding (BARC 3 or 5)

IPD SHARING:
Plan to Share IPD: No